CLINICAL TRIAL: NCT00100334
Title: Multiple Dose Safety and Preliminary Pharmacodynamic Study of PPI-1019 in Subjects With Mild-Moderate Alzheimer's Disease
Brief Title: Safety Study of PPI-1019 in Subjects With Mild-Moderate Alzheimer's Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: PRAECIS Pharmaceuticals Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1019-04-01
Record Dates: First submitted 2004-12-29; First posted 2004-12-30 (Estimated); Last update posted 2006-09-19 (Estimated); Status verified 2006-09

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

INTERVENTIONS:
Drug: PPI-1019 (APAN)

SUMMARY:
This is a single-center, double-blind, inpatient study followed by an outpatient, placebo-controlled, multiple-IV injection evaluation of the safety and tolerability of PPI-1019 in subjects with mild-moderate Alzheimer's disease (AD). The primary objective of the study is to assess the safety of multiple IV injections of PPI-1019 in subjects with mild-moderate Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

* Subject has the ability to understand the requirements of the study, provide written informed consent, and abide by the requirements of the study. In addition, a member of the subject's family or a legally authorized representative must consent to the subject's participation in the study.
* Subject has a caregiver willing to assist the subject's involvement in the study.
* Subject is a male or female between the ages of 50 and 80 with a body mass index (BMI) below 31. Females must be post-menopausal at least 1 year or surgically sterilized.
* Subject must have a cognitive deficit present for at least 1 year and meet DSM -IV criteria for Alzheimer's disease and meet National Institute of Neurological and Communicative Disorders and Stroke/Alzheimer's Disease and Related Disorders Association (NINCDS/ADRDA) criteria for the presence of probable Alzheimer's disease.
* Subject's severity of Alzheimer's disease must be mild-moderate, documented with a Mini Mental State Exam (MMSE) score of 12-26.
* Subject has a computerized tomography (CT) scan or magnetic resonance imaging (MRI) within the prior 12 months which is compatible with a diagnosis of probable AD.
* If a subject is being treated for Alzheimer's disease, it must be with a single cholinesterase inhibitor (donepezil, rivastigmine, or galantamine), with or without memantine, and with a dose which has been stable for at least 3 months prior to dosing.
* Subject performance status is ≤ 3 on items 1 through 5 and ≤ 2 on item 6 from the Degree of Disability Section of the "Rapid Disability Scale-2"
* Subject agrees not to donate blood or blood products while participating in this study and for at least 60 days after discontinuing from the study.

Exclusion Criteria:

* Subject has participated in a clinical trial of another investigational drug or device, or has taken any experimental drug within 30 days prior to admission to the Phase 1 unit. (Subjects previously enrolled in 1019-03-01 may be enrolled in 1019-04-01, only after a wash-out period of 45 days.)
* Subject has a history compatible with vascular dementia as evidenced by a score of 5 or greater on the modified Hachinski Ischemia Scale.
* Subject has evidence of clinically significant unstable cardiovascular, renal, hepatic, gastrointestinal, neurological, or metabolic disease within the past 6 months (as determined by medical history, ECG results, chest x-ray, or physical examination).
* Subject performance status is > 3 on items 1 through 5 and > 2 on item 6 from the Degree of Disability Section of the "Rapid Disability Scale-2."
* Subject has diabetes that requires oral antidiabetic therapy or insulin.
* Subject has a systolic blood pressure (sitting) of greater than 160 mmHg, a diastolic (sitting) greater than 95 mmHg, a decrease in systolic blood pressure of more than 30 mmHg upon standing for 2 minutes from a sitting or supine position, a pulse (sitting or supine) less than 50 or greater than 85.
* Subject has any visual, hearing, or communication disabilities impairing his/her ability to participate in the study.
* Subject is being treated with anticholinergics and/or clinically relevant cytochrome P450 3A4 inducers/inhibitors. The use of other concomitant medications for stable medical conditions is acceptable provided drug and dosage are stable for at least 4 weeks prior to dosing.
* Subject is currently taking herbal supplements which interfere with drug metabolism, e.g. St. John's wort, ginkgo biloba.
* Subject has tested positive for drugs of abuse (amphetamines, barbiturates, cocaine, phencyclidine, or cannabinoids) on screening or Day -1
* Subject has a current or past medical history of alcohol abuse.
* Subject has any elevations (> 1.2 x ULN) on screening or Day -1 for ALT, AST, bilirubin, creatinine, blood urea nitrogen, or alkaline phosphatase.
* Subject has any other screening or Day -1 laboratory values outside the normal ranges that are deemed clinically significant by the investigator.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24
Dates: Start 2004-12; Study Completion 2005-08

PRIMARY OUTCOMES:
Safety will be assessed through the occurrence of clinical adverse events and the occurrence of clinically significant changes from baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Silverado Senior Living, San Juan Capistrano, California, United States